CLINICAL TRIAL: NCT03463382
Title: Erector Spinae Plane Block Versus Quadratus Lumborum Block for Postoperative Analgesia in Children Undergoing Low Abdominal Surgery: A Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block Versus Quadratus Lumborum Block for Postoperative Analgesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Can AKSU, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-95
Record Dates: First submitted 2018-02-28; First posted 2018-03-13 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Pain
Keywords: Pediatric Surgery; Postoperative Pain; Erector spinae plane block; quadratus lumborum block
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP Group (Active Comparator): Erector Spinae Plane Block Group
  Block Drug: 0,25% bupivacaine 0,5ml/kg (max.20ml) were used for blocks
  Interventions: Procedure: Erector Spinae Plane Block; Drug: Bupivacaine (Block Drug)
- QLB Group (Active Comparator): Quadratus Lumborum Block Group
  Block Drug: 0,25% bupivacaine 0,5ml/kg (max.20ml) were used for blocks
  Interventions: Procedure: Quadratus Lumborum Block; Drug: Bupivacaine (Block Drug)

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Erector Spinae Plane block will be administered under general anesthesia before the surgery
  Arms: ESP Group
Procedure: Quadratus Lumborum Block — Quadratus Lumborum Block will be administered under general anesthesia before the surgery
  Arms: QLB Group
Drug: Bupivacaine (Block Drug) — 0,25% Bupivacaine was used 0,5ml/kg (max. 20cc) for block performances

SUMMARY:
Postoperative pain management in children is still standing as a problem to solve. Effect of quadratus lumborum block has been shown to be a promising technique to overcome postoperative pain in children undergoing low abdominal surgeries. Erector spinae plane block is a new defined relatively safer and easier regional anesthesia technique which could be used for this purpose. Primary aim of this double blinded randomized controlled trial is to compare the analgesic efficacy of this two block techniques in this group of pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* 1-7 years of age
* ASA I-II
* Undergoing elective low abdominal surgery

Exclusion Criteria:

* infection of the skin at the site of needle puncture area
* patients with known allergies to any of the study drugs
* coagulopathy
* ASA III-IV
* Patients with neurological disorders

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Pain scores | Postoperative first 6hours
  FLACC scale will be used. The Face, Legs, Activity, Cry, Consolability scale or FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.

SECONDARY OUTCOMES:
Time to first analgesic drug | first 48 hour
  Time to first analgesic drug will be recorded
Need for analgesic | 24 hour
  Number of patients who required analgesic in the first 24 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Hospital, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aksu C, Sen MC, Akay MA, Baydemir C, Gurkan Y. Erector Spinae Plane Block vs Quadratus Lumborum Block for pediatric lower abdominal surgery: A double blinded, prospective, and randomized trial. J Clin Anesth. 2019 Nov;57:24-28. doi: 10.1016/j.jclinane.2019.03.006. Epub 2019 Mar 6. PMID 30851499